CLINICAL TRIAL: NCT03698526
Title: Virtual Reality for Symptoms Control in Palliative Care
Acronym: VRPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Palliativnetz Muenster gGmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: VRPC2018
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Palliative Care; Virtual Reality; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Palliative care I (Active Comparator): Palliative care
  Interventions: Device: Samsung Gear VR, Galaxy S8, Applied VR App
- Control II (Active Comparator): Patients with mamma carcinoma and (neo-) adjuvant radiotherapy
  Interventions: Device: Samsung Gear VR, Galaxy S8, Applied VR App
- Control III (Active Comparator): Patients before colonoscopy
  Interventions: Device: Samsung Gear VR, Galaxy S8, Applied VR App

INTERVENTIONS:
Device: Samsung Gear VR, Galaxy S8, Applied VR App — Virtual Reality Experience

SUMMARY:
The aim of this study is to evaluate how Virtual Reality (VR) can be used to control symptoms and improve the quality of life in palliative care. The interventional prospective case control study is planned to contain five phases including two control groups. The following describes only phase one to three.

In the pilot phase patients get a one-time application of the VR-Technology. After that, two control groups will be recruited from patients with 1. mamma carcinoma and the indication of (neo-) adjuvant radiotherapy and 2. before a colonoscopy-treatment. Both groups receive the VR application before treatment (radiotherapy/colonoscopy).

This first part proofs the application of Virtual Reality on patients in palliative care with the aim to control symptoms and reduce pain and anxiety.

The clinical study hypothesis bases on the assumption that VR reduces pain and anxiety and may have a positive influence on their quality of life.

DETAILED DESCRIPTION:
Pilot phase:

After the enrolment and consent of participation the patient receives a questionnaire consisting of different independent assessments. The visual analogue scale with values from 1 to 10 quantifies subjective pain. A functional pain questionnaire (Pain-Out) is developed to assess the pain in between the last seven days, the associated limitations, the actions and side effects of combined pain therapy.

To measure the generic health-related quality of life the patient is asked to answer the EuroQoL Group 5-Dimension 5-Level Self Report Questionnaire (EQ-5D-5L).

A Virtual Reality application is offered immediately after the questionnaire has been completed. Following the application of VR the patient will receive VAS and functional pain questionnaires again to assess the change from baseline.

Control phase:

The following control phase is to review the effectiveness of VR application on the basis of two different control groups. In a randomized setting 30 patients with mamma carcinoma receive an application of VR before their radiotherapy. The second control group consists of 40 patients with an individual indication of a colonoscopy.

Instead of pain by VAS and QoL in the pilot phase each patient receives now the Hospital Anxiety and Depression Scale (HADS) before and after the application. The Functional Pain Questionnaire remains with the control group of patients with mamma carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Patient understands information for participation
* Patients are able to give informed written consent
* (Informed written) consent prior inclusion in study
* study arm I: Indication for palliative care due to any advanced life-limiting and progressive diseases
* control II: Patients with mamma carcinoma and (neo-) adjuvant radiotherapy
* control III: Patients before colonoscopy

Exclusion Criteria:

* Epileptic seizures in medical history
* Patients with claustrophobia
* Patients with tendency to vertigo and motion sickness
* Age under 18 years
* No informed written consent
* Inability to understand information for participation, language difficulties (foreign nationals), hardness of hearing
* Blindness

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Pain by VAS | peri-interventional
  Pain by VAS (visual analogue scale), Pain is indicated on a 100mm visual scale, the patient can report no pain (0 mm) to maximum pain (100mm).
Hospital Anxiety and Depression Scale | peri-interventional
  Hospital Anxiety and Depression Scale, Questionnaire to indicate anxiety and depression, 14 questions (7 depression, 7 anxiety) with 4 possibilities to answer, validated questionnaire according to Zigmond et al. (Zigmond, A. S. & Snaith, R. P. The hospital anxiety and depression scale. Acta psychiatrica Scandinavica 67, 361-370 (1983))

SECONDARY OUTCOMES:
Functional pain by Pain-Out-Questionnaire | peri-interventional
  Functional pain by Pain-Out-Questionnaire, Questionnaire in which the patient can indicate pain according to functionality (physical activity, sleeping, breathing) and feeling associated to pain (helplessness, nausea, drowsiness, Pruritus, diszziness), Scales from 0 (no symptom) to 10 (intense).
Quality of life by EQ-5D-5L | peri-interventional
  Quality of life by EQ-5D-5L, 5 Items Questionnaire and Scale from 0 (worst health status) to 100 (perfect health status), indicated by the patients, validated questionnaire according to Hinz et al. (Hinz, A., Kohlmann, T., Stobel-Richter, Y., Zenger, M. & Brahler, E. The quality of life questionnaire EQ-5D-5L: psychometric properties and normative values for the general German population. Quality of life research : an international journal of quality of life aspects of treatment, care and rehabilitation 23, 443-447, doi:10.1007/s11136-013-0498-2 (2014).)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Lenz, MD, Principal Investigator — Institut of Palliative Care, University Hospital of Muenster
Locations (2):
- Germany (2):
  - Palliativnetz Muenster gGmbH, Münster, North Rhine-Westphalia
  - University Hospital Muenster, Münster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teunissen SC, Wesker W, Kruitwagen C, de Haes HC, Voest EE, de Graeff A. Symptom prevalence in patients with incurable cancer: a systematic review. J Pain Symptom Manage. 2007 Jul;34(1):94-104. doi: 10.1016/j.jpainsymman.2006.10.015. Epub 2007 May 23. PMID 17509812
- [Background] Gold JI, Mahrer NE. Is Virtual Reality Ready for Prime Time in the Medical Space? A Randomized Control Trial of Pediatric Virtual Reality for Acute Procedural Pain Management. J Pediatr Psychol. 2018 Apr 1;43(3):266-275. doi: 10.1093/jpepsy/jsx129. PMID 29053848
- [Background] Mosadeghi S, Reid MW, Martinez B, Rosen BT, Spiegel BM. Feasibility of an Immersive Virtual Reality Intervention for Hospitalized Patients: An Observational Cohort Study. JMIR Ment Health. 2016 Jun 27;3(2):e28. doi: 10.2196/mental.5801. PMID 27349654
- [Background] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- [Background] Hoffman HG, Patterson DR, Carrougher GJ, Sharar SR. Effectiveness of virtual reality-based pain control with multiple treatments. Clin J Pain. 2001 Sep;17(3):229-35. doi: 10.1097/00002508-200109000-00007. PMID 11587113